CLINICAL TRIAL: NCT07005830
Title: Examining the Impact of a Specific Guided Meditation (Twin Hearts Meditation; THM) on Mood, Cognitive Functioning, and EEG Dynamics in Experienced and Novice Meditators
Brief Title: The Impact of Twin Hearts Meditation on Mood, Cognitive Functioning, and EEG Dynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroMeditation Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024-0250
Record Dates: First submitted 2025-04-17; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Positive Mood States; Negative Mood States; Cognitive Processing Speed; Cognitive Flexibility
Keywords: meditation; Electroencephalography; emotional regulation; Trail Making Test; Cognitive Neuroscience; mood; P300
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Unblinded control group comparison (2x2 factorial design) with multi-modal measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Impact of Meditation on Mood, Cognitive Function, & EEG Dynamics by Meditation Experience Level (Experimental): Twin Hearts Meditation (THM) is a 21-minute guided meditation practice developed by Master Choa Kok Sui as part of Pranic Healing & Arhatic Yoga (Sui, 2005). It is designed to promote spiritual development, emotional balance, and cognitive well-being by activating and harmonizing the heart chakra (emotional love) and the crown chakra (divine love and higher consciousness). The meditation is based on the principle that blessing the Earth with loving-kindness leads to inner transformation and heightened awareness. The meditation itself is divided into several sections that include (in order of appearance), an invocation for divine blessings, an abbreviated prayer of St. Francis of Assisi, activation of the heart and crown chakras, blessing the Earth with lovingkindness, chanting the mantra "OM," silent meditation, and a closing.
  Interventions: Behavioral: Twin Hearts Meditation

INTERVENTIONS:
Behavioral: Twin Hearts Meditation — Twin Hearts Meditation (THM) is a 21-minute guided meditation practice developed by Master Choa Kok Sui as part of Pranic Healing & Arhatic Yoga (Sui, 2005).

SUMMARY:
The goal of this clinical trial is to examine the impact of a specific guided meditation (Twin Hearts Meditation; THM) on cognitive functioning and EEG dynamics in experienced and inexperienced meditators.

The main questions it aims to answer are:

* Will the experienced meditators outperform inexperienced meditators on the attention control tasks (Flanker, Trails A & B) at baseline (pre-meditation)?
* Will both groups show improvements in performance after meditation associated with mood and physiological state changes?
* Will the experienced meditators show an overall mood profile of higher positive mood states and less negative mood states (Brunel Mood Scale subscale difference) at baseline (pre-meditation)?
* Will both groups show mood state improvements after meditation?
* Will the experienced meditators show differences in electrophysiological characteristics compared to inexperienced meditators?
* Will inexperienced meditators exhibit shifts from their baseline resting-state EEG towards being more similar to the EEG characteristics of experienced meditators at baseline?
* Will experienced meditators demonstrate differences in P300 latencies and amplitudes on the auditory oddball paradigm.

Participants will:

* Take a series of pre-meditation surveys.
* Complete pre-meditation P300 auditory oddball task.
* Complete pre-meditation cognitive behavioral task set.
* Continuous 19-channel EEG recording before and after pre-recorded guided THM.
* Take a series of post-meditation surveys.
* Complete post-session P300 auditory oddball task.
* Complete post-session cognitive behavioral task set.

DETAILED DESCRIPTION:
Eighteen experienced Arhatic Yoga practitioners and 18 novice meditators were recruited for this study. Experienced meditators were recruited from a weeklong Arhatic Yoga Spiritual Retreat (July 20-28, 2024) in Bovina, NY. Inclusion to the experienced meditator sample included a minimum of 1,000 hours practice of THM as well as a current meditation practice. Inexperienced meditators were recruited in Eugene, OR, via social media and community flyers. Inclusion criteria for this sample included less than 10 hours of lifetime meditation practice. Compensation for the inexperienced group was a $30 check or paypal credit.

Screening of inclusion and exclusion criteria was completed via digital forms. Those deemed eligible completed the informed consent process, and provided more demographic information for sample characteristics.

Experimental Design

The experiment was an unblinded, control group comparison (2 x 2 factorial design) of experienced versus novice meditators groups with multimodal measurements (subjective mood questionnaire, cognitive tasks, neural/ EEG) taken before and after completion of a Twin Hearts Meditation practice. Both experienced and meditation naïve subjects underwent a structured research protocol consisting of screening, a pre-meditation assessment, a guided Twin Hearts Meditation session, and a post-meditation assessment. Sessions lasted about 90 min. The procedure was as follows:

Screening and Participant Selection. Participants completed an online screening and demographic questionnaire. Those meeting inclusion and exclusion criteria were invited to participate in the research study. Eligible subjects who indicated interest were scheduled for a laboratory-based session. Informed consent procedures were provided upon arrival to the lab space ahead of conducting the remaining protocol procedures.

Pre-Meditation Assessment. After obtaining informed consent, subjects completed a series of neural, mental and cognitive baseline measures. Psychological questionnaires included the Multidimensional Psychological Flexibility Inventory abbreviated scale (MPFI - Abbreviated Flexibility), and the Tellegen Absorption Scale (to assess baseline mental traits). These two measures were only given once for assessing baseline trait differences between experimental meditator samples. However, the following measures were given before and after meditation:

Participants next completed the Brunel Mood Scale. Then subjects were prepared for EEG to measure neural activity in a 3-minute resting state recording, as well as during their completion of a P300 auditory oddball task. They then completed the cognitive-behavioural task set, that included the Flanker task (to evaluate response inhibition and attention control) and Trail Making Tests A (to assess processing speed, simple attention) & B (complex attention/executive function).

Twin Hearts Meditation Session. Participants then listened to a pre-recorded 21-minute guided Twin Hearts Meditation session via headphones with eyes closed. Participants were instructed to simply follow along with the instructions provided in the meditation.

Post-Meditation Assessment. Following the meditation, subjects completed the post-meditation EEG baseline recording. Additional mental given: i ) Depth of Meditation Scale (to assess subjective meditation experience), ii) Brunel Mood Scale (to measure post-meditation mood state). This was followed by re-administration of the Cognitive-Behavioural measurement tasks (P300 auditory oddball, Flanker, Trail Making Test A & B)

Description of Psychological Questionnaire-based Measurements

Demographic questionnaire. This survey asks basic questions regarding age, sex, history of mental health diagnoses, and meditation history. Data was used from this survey to characterize overall and Experienced versus Inexperienced meditator sample characteristics.

Tellegren Absorption Scale (TAS). The Tellegen Absorption Scale is a 34-item multi-dimensional measure that assesses imaginative involvement and the tendency to become mentally absorbed in everyday tasks. Each item on the scale requires a 'true' or 'false' response. Scores for the TAS and its subscales reflect the number of questions marked 'true,' with higher scores indicating higher absorption. Tellegen reported an internal reliability of .88 and a 30-day test-retest reliability of .91. Kihlstrom reported a test-retest reliability of .85.

The TAS is divided into five subscales: altered states of consciousness (TAS-ACS; "I sometimes 'step outside' my usual self and experience an entirely different state of being"), aesthetic involvement in nature (TAS-AIN; "I like to watch cloud shapes change in the sky"), imaginative involvement (TAS-II; "I am able to wander off into my thoughts while doing a routine task and actually forget that I am doing the task, and then find a few minutes later that I have completed it"), Synesthesia (TAS-SYN; "I find that different odors have different colors"), and extrasensory perception or ESP (TAS-ESP; "I can often somehow sense the presence of another person before I actually see her/him"). A high score on a specific subscale indicates a greater tendency to experience that particular type of absorption, with the TAS Total score reflecting an overall trait of responsive absorption to stimuli, tasks, and surroundings.

Psychological Flexibility Scale (PFS). The Psychological Flexibility Scale (PFS) is a shorter global composite of the Multidimensional Psychological Flexibility Inventory. The 12-item PFS is comprised of the first two items of each of the MPFI subscales that subjects respond to using on a six-point Likert scale to rate the accuracy of statement related to acceptance, present moment awareness, self as context, defusion, values, and committed action. Higher scores indicate higher mental flexibility comprised by the item pairs in each domain.

Depth of Meditation Experience. The Meditation Depth Questionnaire is a 30-item self-report measure designed to assess the depth of meditative experience across five progressive stages. These stages include: (1) Hindrances, which captures difficulties such as boredom, impatience, and trouble with concentration (reverse-coded for consistency); (2) Relaxation, reflecting feelings of inner peace and calmness; (3) Concentration, describing detachment from thoughts, deep insight, and mental clarity; (4) Essential Qualities, encompassing emotions like love, gratitude, and connectedness; and (5) Non-Duality, representing the dissolution of cognitive processes and a sense of unity. The questionnaire is given post-meditation to evaluate subjective depth of experience, with higher scores indicating greater meditative depth across individual subscales and overall. The Hindrance scale was reverse coded, to be in line with other scales and total score, so that higher values indicate more favorable experiences overall and according to subscales.

Brunel Mood Scale. The Brunel Mood Scale is a 32-item self-report measure designed to assess current mood states. It consists of eight unipolar mood dimensions: anger, tension, depression, vigor, fatigue, confusion, happiness, and calmness. Participants respond to the prompt, "How do you feel right now?" by rating each mood descriptor on a 5-point Likert scale (0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, 4 = extremely), indicating the intensity of their momentary emotional experience. As well as producing subscale scores, an overall mood score, referred to as a Total Mood Disturbance (TMD) score, can be calculated by summing the scores for Tension, Depression, Anger, Fatigue and Confusion and then subtracting the Vigor score. Higher TMD scores indicate greater overall mood disturbance, reflecting higher levels of negative emotions inversely correlated with lower positive affect. Conversely, lower scores suggest better mood balance and emotional well-being.

Description of Cognitive-Behavioral Measures

Trails A & B. Trails A & B is a cognitive assessment measurement consisting of two tasks, Trail A and Trail B. Trail A measures visual processing speed and simple attention, requiring subjects to connect numbers in sequential order across a display sheet. For Trail B subjects must complete a task similar to Trail A, but instead alternate between numbers and letters intermixed across the display, in ascending order. Trail B is considered a measure of complex attention and working memory, and of executive function including inhibition and divided attention. Trails A & B were given digitally using the WAVi Software Platform under the supervision of a researcher. Instructions were provided via computer and researcher. Performance metrics included the number o

Statistical Analysis Statistical analyses were conducted using SPSS. Prior to hypothesis testing, data were screened for missing values, outliers, normality, and homogeneity of variance assumptions. Variables were evaluated for normality evaluating for skewness and kurtosis values between +2/-2 and +7/-7 respectively. Levene's tests of homogeneity were also conducted, p < 0.05. A combination of ANOVA, t-testing, and correlational analyses were used for hypothesis testing. All statistical tests were two-tailed, with an alpha level set at .05. Effect sizes and 95% confidence intervals (±1.96 SEM) are reported where appropriate.

The primary approach for hypothesis testing involved running 2 (Experimental Group: Experienced, Inexperienced) X 2 (Time: Pre-meditation, Post-meditation) repeated-measures ANOVAs (rm-ANOVA) for the Brunel Mood Scale, Flanker performance measures, Trails A&B performance measures, P300 and Resting state EEG measures of interest. The stepwise Holm-Bonferroni correction (Holm, 1979) was applied to control for family-wise error of questionnaire, cognitive/attentional task, and EEG variable sets initially investigated by ANOVA sets, and applied for follow-up on pairwise comparisons where significant interaction effects were found.

One-way ANOVA and independent t-tests were used to investigate demographic, baseline and single time point comparisons between groups (e.g., TAS, depth of meditation experience). Chi-Square testing was conducted for applicable frequency-based values of the demographic variables.

In addition, Pearson's correlation analyses were conducted in planned and ad hoc approaches. Planned correlations included [ ]. Unplanned/exploratory correlations included assessing the relationship of variables discovered to be statistically significant in ANOVA results, with other variables that might help further describe or inform interpretation of a result. Correlation coefficients were interpreted following Cohen's guidelines, where values of 0.10, 0.30, and 0.50 were considered small, medium, and large, respectively. To control for multiple comparisons, a Benjamini-Hochberg false discovery rate (FDR) correction was applied (I have not yet applied this and may not - need specified correlation sets before deciding)

Data Cleaning and Outlier Handling Outlier detection was performed using a combination of visual inspection (boxplots, Q-Q plots), and statistical thresholds (interquartile method). Extreme outliers were removed as single data points, or winzored with imputation. The decision for complete omission versus imputation was dependent on the type and amount of missing or omitted data. Imputation was selectively and sparingly used for resting state EEG, whereby unrealistic outlier values (suspected of being artefact, missed on built-in software filtering and cleaning) were removed, then re-estimated with regression imputation based on group-time point averages and proximal electrode site values.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* English speaking
* capable of providing consent.

Exclusion Criteria:

- history of traumatic brain injury or serious mental health concerns (schizophrenia, bipolar disorder)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-07-21 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Mood Differences and Changes in Experienced vs. Inexperienced Meditators | the 25 minutes of the pre-recorded meditation
  This study examines both baseline mood differences & post-meditation mood changes between experienced & inexperienced meditators using Brunel Mood Scale, a 32-item self-report measure designed to assess current mood states. It consists of 8 unipolar mood dimensions: anger, tension, depression, vigor, fatigue, confusion, happiness & calmness. Participants respond to prompt "How do you feel right now?" by rating each mood descriptor on a 5-point Likert scale (0=not at all to 4=extremely), indicating intensity of their momentary emotional experience. As well as producing subscale scores, an overall Total Mood Disturbance (TMD) score can be calculated by summing the scores for Tension, Depression, Anger, Fatigue & Confusion and then subtracting Vigor score. Higher TMD scores indicate greater overall mood disturbance, reflecting higher levels of negative emotions inversely correlated with lower positive affect. Conversely, lower scores suggest better mood balance & emotional well-being.
Cognitive Performance in Experienced vs. Inexperienced Meditators: Trail Making A Outcomes | 5 minutes
  This study examines cognitive changes using the Trail Making Test-A (TMT-A), which assesses processing speed (TMT-A) by measuring the time taken to connect a sequence of numbers. Performance metrics included the number of errors per trial and time to completion, with the latter serving as the primary performance indicator.
Cognitive Performance in Experienced vs. Inexperienced Meditators: Trail Making B Outcomes | 5 minutes
  This study examines cognitive changes using the Trail Making Test-B (TMT-B) which assesses cognitive flexibility/executive function (TMT-B) by measuring the time taken to connect a sequence of alternating numbers and letters. Performance metrics included the number of errors per trial and time to completion, with the latter serving as the primary performance indicator.
Cognitive Performance in Experienced vs. Inexperienced Meditators: Flanker Test Selective Attention Outcomes | 5 minutes
  This study examines cognitive changes using the Flanker Test. Participants are required to quickly identify a central target stimulus while ignoring distracting stimuli on either side, measuring their ability to maintain focus despite interference. In this study, the Flanker Task was administered using the WAVi software platform, with a total test duration of approximately five minutes. Performance metrics include the number of total errors.
Cognitive Performance in Experienced vs. Inexperienced Meditators: Flanker Test Inhibitory Control Outcomes | the 25 minutes of the pre-recorded meditation
  This study examines baseline cognitive differences and post-meditation cognitive changes between experienced and inexperienced meditators using the Flanker Test. The Flanker test evaluates inhibitory control defined as the ability to suppress the influence of the flankers and respond correctly to the control.
  Participants are required to quickly identify a central target stimulus while ignoring distracting stimuli on either side, measuring their ability to maintain focus despite interference. In this study, the Flanker Task was administered using the WAVi software platform, with a total test duration of approximately five minutes. Performance metrics include the error rates for congruent and incongruent flanker trials.
P300 Event-Related Potential in Experienced vs. Inexperienced Meditators: Amplitude Outcomes | the 25 minutes of the pre-recorded meditation
  Study examines baseline neurocognitive differences & post-meditation changes in P300 event-related potentials (ERPs) between experienced & inexperienced meditators, using auditory oddball paradigm to assess amount of cognitive resources used. Task consisted of 200 common tones & 40 randomly presented rare (higher-pitched) tones, at 1 Hz.
  Participants pressed mouse button upon hearing rare tone. Before beginning, participants had opportunities to practice task to ensure comprehension & accuracy. Measurements acquired & used for analyses included p300 amplitude. Higher amplitude indicates more attention was allocated to the stimulus and suggests stronger engagement, better stimulus discrimination, and/or higher motivation.
P300 Event-Related Potential in Experienced vs. Inexperienced Meditators: Latency Outcomes | the 25 minutes of the pre-recorded meditation
  Study examines baseline neurocognitive differences & post-meditation changes in P300 event-related potentials (ERPs) between experienced & inexperienced meditators, using auditory oddball paradigm to assess cognitive efficiency. Task consisted of 200 common tones & 40 randomly presented rare (higher-pitched) tones, at 1 Hz.
  Participants pressed mouse button upon hearing rare tone. Before beginning, participants had opportunities to practice task to ensure comprehension & accuracy. Measurements acquired & used for analyses included p300 latency. Latency refers to the time delay, in milliseconds, between presentation of a target stimulus and peak of the P300 wave. It reflects the speed of stimulus evaluation & decision-making processes. Shorter P300 latencies indicate faster cognitive processing, whereas longer latencies are associated with delayed neural responses, often observed in people with cognitive impairments or attentional deficits.
Alpha Peak Frequency in Experienced vs. Inexperienced Meditators | the 25 minutes of the pre-recorded meditation
  This study examines baseline neurophysiological differences and post-meditation changes alpha peak frequency (APF) between experienced and inexperienced meditators.
  Alpha Peak Frequency (APF): Reflects the speed of intrinsic neural oscillations, with higher APF linked to greater cognitive efficiency, attentional stability, and mental flexibility.
Frontal Asymmetry in Experienced vs. Inexperienced Meditators | the 25 minutes of the pre-recorded meditation
  This study examines baseline neurophysiological differences and post-meditation changes in EEG frontal asymmetry, between experienced and inexperienced meditators. These measures provide insights into cognitive flexibility, attentional control, emotional regulation, and meditation-induced neural adaptations.
  Frontal Alpha Asymmetry (FAA): Measures relative left vs. right frontal alpha power, where greater rightward asymmetry is associated with approach motivation and positive affect, while leftward asymmetry is linked to withdrawal tendencies and negative mood.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Viczko, PhD, Study Director
Locations (1):
- NeuroMeditation Institute, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zeidan F, Johnson SK, Diamond BJ, David Z, Goolkasian P. Mindfulness meditation improves cognition: evidence of brief mental training. Conscious Cogn. 2010 Jun;19(2):597-605. doi: 10.1016/j.concog.2010.03.014. Epub 2010 Apr 3. PMID 20363650
- [Background] Travis F, Haaga DA, Hagelin J, Tanner M, Arenander A, Nidich S, Gaylord-King C, Grosswald S, Rainforth M, Schneider RH. A self-referential default brain state: patterns of coherence, power, and eLORETA sources during eyes-closed rest and Transcendental Meditation practice. Cogn Process. 2010 Feb;11(1):21-30. doi: 10.1007/s10339-009-0343-2. Epub 2009 Oct 28. PMID 19862565
- [Background] Tellegen A, Atkinson G. Openness to absorbing and self-altering experiences ("absorption"), a trait related to hypnotic susceptibility. J Abnorm Psychol. 1974 Jun;83(3):268-77. doi: 10.1037/h0036681. No abstract available. PMID 4844914
- [Background] Tarrant JM, Raines N, Blinne WR. The Effects of Meditation on Twin Hearts on P300 Values: A Repeated Measures Comparison of Nonmeditators and the Experienced. Integr Med (Encinitas). 2019 Apr;18(2):36-41. PMID 31341443
- [Background] Lan MF, Lane AM, Roy J, Hanin NA. Validity of the Brunel Mood Scale for use With Malaysian Athletes. J Sports Sci Med. 2012 Mar 1;11(1):131-5. eCollection 2012. PMID 24149128
- [Background] Singhal, T., Manjhi, D., & Kumar, S. (2015). Neuroplastic changes following Twin Hearts Meditation: A functional MRI study. Indian Journal of Psychiatry, 57(3), 281-286.
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Background] Rolffs JL, Rogge RD, Wilson KG. Disentangling Components of Flexibility via the Hexaflex Model: Development and Validation of the Multidimensional Psychological Flexibility Inventory (MPFI). Assessment. 2018 Jun;25(4):458-482. doi: 10.1177/1073191116645905. Epub 2016 May 5. PMID 27152011
- [Background] Mrazek MD, Franklin MS, Phillips DT, Baird B, Schooler JW. Mindfulness training improves working memory capacity and GRE performance while reducing mind wandering. Psychol Sci. 2013 May;24(5):776-81. doi: 10.1177/0956797612459659. Epub 2013 Mar 28. PMID 23538911
- [Background] Leiberg S, Klimecki O, Singer T. Short-term compassion training increases prosocial behavior in a newly developed prosocial game. PLoS One. 2011 Mar 9;6(3):e17798. doi: 10.1371/journal.pone.0017798. PMID 21408020
- [Background] Lehrer P, Kaur K, Sharma A, Shah K, Huseby R, Bhavsar J, Sgobba P, Zhang Y. Heart Rate Variability Biofeedback Improves Emotional and Physical Health and Performance: A Systematic Review and Meta Analysis. Appl Psychophysiol Biofeedback. 2020 Sep;45(3):109-129. doi: 10.1007/s10484-020-09466-z. PMID 32385728
- [Background] Hutcherson CA, Seppala EM, Gross JJ. Loving-kindness meditation increases social connectedness. Emotion. 2008 Oct;8(5):720-4. doi: 10.1037/a0013237. PMID 18837623
- [Background] Holm, S. (1979). A Simple Sequentially Rejective Multiple Test Procedure. Scand. J. Stat. 6 (2), 65-70.
- [Background] Fox KC, Nijeboer S, Dixon ML, Floman JL, Ellamil M, Rumak SP, Sedlmeier P, Christoff K. Is meditation associated with altered brain structure? A systematic review and meta-analysis of morphometric neuroimaging in meditation practitioners. Neurosci Biobehav Rev. 2014 Jun;43:48-73. doi: 10.1016/j.neubiorev.2014.03.016. Epub 2014 Apr 3. PMID 24705269
- [Background] Farb NA, Segal ZV, Mayberg H, Bean J, McKeon D, Fatima Z, Anderson AK. Attending to the present: mindfulness meditation reveals distinct neural modes of self-reference. Soc Cogn Affect Neurosci. 2007 Dec;2(4):313-22. doi: 10.1093/scan/nsm030. PMID 18985137
- [Background] Chambers, R., Lo, B. C., & Allen, N. B. (2008). The impact of intensive mindfulness training on attentional control, cognitive style, and affect. Cognitive Therapy and Research, 32(3), 303-322.
- [Background] Alexander CN, Langer EJ, Newman RI, Chandler HM, Davies JL. Transcendental meditation, mindfulness, and longevity: an experimental study with the elderly. J Pers Soc Psychol. 1989 Dec;57(6):950-64. doi: 10.1037//0022-3514.57.6.950. PMID 2693686